CLINICAL TRIAL: NCT05638984
Title: A Low Dose Decitabine Combined With Tirelizumab Prospective Phase II Clinical Study Comparing Tirelizumab in Patients With Advanced Esophageal Squamous Cell Carcinoma Who Did Not Progress With First-line Immunotherapy Combined With Chemotherapy
Brief Title: Low Dose Decitabine in Combination With Tirelizumab Comparison of Tirelizumab in the First-line Treatment of Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu hui, associate senior doctor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-IIT-001
Record Dates: First submitted 2022-11-16; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: PFS
MeSH Terms: interventions — Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose decitabine combined with tirelizumab (Experimental): Injection site citabine, 10 mg/ bottle, 10 mg/d, Q3W, D1-D5 intravenous infusion; Tirelizumab injection 200mg D5 intravenous infusion.
  Interventions: Drug: Decitabine Injection; Drug: tirelizumab
- tirelizumab (Active Comparator): Tirelizumab injection, 10ml: 100mg/1 bottle, 200mg, Q3W, D1 IV infusion.
  Interventions: Drug: tirelizumab

INTERVENTIONS:
Drug: Decitabine Injection — Injection site citabine, 10 mg/ bottle, 10 mg/d, Q3W, D1-D5 intravenous infusion; Tirelizumab injection 200mg D5 intravenous infusion
  Other Names: tirelizumab
  Arms: low-dose decitabine combined with tirelizumab
Drug: tirelizumab — 10ml: 100mg / 1 bottle, 200mg, Q3W, D1 i. v. infusion.

SUMMARY:
To evaluate the efficacy and safety of low-dose decitabine combined with tirelizumab in the treatment of patients with advanced esophageal squamous cell carcinoma who did not progress in first-line immunotherapy combined with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects voluntarily participate and sign written informed consent; Age ≥18 years; Confirmed by histopathology and/or cytology as esophageal squamous cell carcinoma; At least one measurable lesion according to AJCC 8th staging and RECIST 1.1 solid tumor evaluation criteria.

Those who have received immunocheckpoint inhibitors combined with chemotherapy (e.g., paclitaxel + cisplatin) in the first line, and the disease has not progressed;

Good functioning of major organs, no serious uncontrolled hypertension, diabetes and heart disease, that is, the relevant indicators within 14 days before treatment meet the following requirements:

* ANC≥1.2×109/L and lymphocyte count ≥0.5×109/L without the support of granulocyte colony stimulating factor;
* Without blood transfusion, patients with platelet count ≥100×109/L and hemoglobin ≥90g/L can meet the criteria through blood transfusion;
* AST, ALT and ALP≤2.5× upper limit of normal (ULN), total bile red ≤1.5×ULN, except the following conditions: for known Gilbert patients: total bilirubin ≤3×ULN, creatinine ≤1.5×ULN, albumin ≥25g/L;
* For patients not receiving anticoagulant therapy: INR and aPTT≤1.5×ULN. estimated survival ≥3 months; Score of ECOG physical strength: 0~1; The ability of patients to follow the study protocol according to the judgment of the investigator.

Exclusion Criteria:

Previous immunotherapy; no measurable lesions; There are small cell carcinoma, adenocarcinoma or mixed carcinoma components in the histology; Complete esophageal obstruction; Any NCI CTCAE≥ Grade 2 toxicity that has not recovered after previous chemotherapy; High risk of esophageal fistula was found through clinical evaluation or imaging examination, such as history of esophageal fistula or related symptoms, or primary tumor infiltration into large blood vessels or trachea; had positive detection for EB virus (EBV) capsid antigen IgM during screening (PCR method); If a patient requires analgesic treatment, the treatment regimen used at the time of enrollment must be stable; The men who have HIV positive results at the time of screening; people who test positive for hepatitis C virus (HCV) during sieving; HBV positive screening, and cccDNA≥500 IU/mL; Any of the following diseases in the 12 months prior to enrollment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, or cerebrovascular accident; Pregnant or lactating women or fertile but did not take contraceptive measures; suffer any other serious physical or mental problem of an acute or chronic nature; judging by the researchers, that doesn't fit to participate in the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | At the end of last Cycle (each cycle is 21 days)
  Progression-Free Survival